CLINICAL TRIAL: NCT02994160
Title: DExterous Hand Control Through Fascicular Targeting (DEFT) - (Human Subjects)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Defense Advanced Research Projects Agency (U.S. Federal Agency); Nerves Incorporated, Inc. (Unknown); Arizona State University (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Jonathan Cheng, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU 092014-061
Record Dates: First submitted 2016-12-12; First posted 2016-12-15 (Estimated); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Amputation; Traumatic, Hand
Keywords: peripheral nerve; intraneural electrode; hand amputation; forearm amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- Fast electrodes (Experimental): Implant temporary Fast electrodes and record the nerve signals that control delicate finger motions and play back the nerve signals that give the hand feelings of touch and movement.
  Interventions: Other: Fast electrode

INTERVENTIONS:
Other: Fast electrode — Implant temporary Fast electrodes and record the nerve signals that control delicate finger motions and play back the nerve signals that give the hand feelings of touch and movement.

SUMMARY:
Our goal is to temporarily implant the following groups for 540 +/- 30 days:

1. Forearm FAST electrodes

   1. Five human partial hand amputees (amputated at the level of the hand) with 2 FAST electrodes in the ulnar nerve and 2-5 FAST electrodes in the median nerve.
   2. Five human hand and forearm amputees (amputated at the level of the forearm) with 2 FAST electrodes in the ulnar nerve and 2-5 FAST electrodes in the median nerve .
2. Arm FAST electrodes

   1. Five human partial hand amputees (amputated at the level of the hand) with 2 FAST electrodes in the ulnar nerve and 2-5 FAST electrodes in the median nerve.
   2. Five human hand and forearm amputees (amputated at the level of the forearm) with 2 FAST electrodes in the ulnar nerve and 2-5 FAST electrodes in the median nerve.
   3. Five human hand, forearm and arm amputees (amputated at the level of the arm) with 2 FAST electrodes in the ulnar nerve and 2-5 FAST electrodes in the median nerve.

DETAILED DESCRIPTION:
Study Procedures:

Subjects will be consented during a pre-operative visit in the Plastic Surgery Clinic and screened for participation.

Screening history and physical Potential human subjects will receive a full medical assessment by the PI. The screening interview will focus on details of the patient's upper extremity condition and comprehensive details of the patient's overall health status. The screening examination will include general examination of the subject.

Pre-operative imaging and diagnostic studies MRI, x-ray, EMG/Nerve conduction studies (NCS) - Each subject who passes the screening H&P will receive the following for their residual limb: magnetic resonance neurogram (MRN), plain x-rays, EMG/nerve conduction studies, and psychological assessment. Other studies will be performed in accordance with the UT (University of Texas) Southwestern pre-operative testing protocol, and will depend on the age/gender/medical history of the subject.

MR neurogram will provide information regarding the location and health of amputated peripheral nerve stumps in the residual limb.

Plain x-rays will allow assessment of the bony anatomy of the amputation stump, and suitability for nerve/muscle implants.

Electromyogram/Nerve conduction studies will include motor and sensory nerve conduction of the median and ulnar nerves, and needle exam (voluntary activation EMG) of the residual arm, forearm and hand muscles.

A comprehensive assessment will be completed by a licensed psychologist. This assessment is utilized to ensure that patient is psychologically and mentally suitable to participate in the study.

Other studies Based on UT Southwestern pre-operative testing protocol, other studies may be required prior to surgery. CBC (complete blood count) with type and screen will be performed, and HCG (pregnancy test) in females age 15-50. EKG will be performed in males > 40, and females > 50. Chest x-ray will be performed in subjects with a prior history of smoking or lung/chest injury. If surgery is scheduled for more than 90 days after this testing is completed, another set of tests will be needed.

Patient treatment, week of surgery Subjects who have passed all screening measures and who have completed the consent process will be seen for a routine pre-operative H&P up to 30 days before surgery.

Prophylaxis for Methicillin-Resistant Staph Aureus (MRSA) The subject will receive mupirocin ointment to place intranasal, to both nares, twice a day for 5 days prior to surgery.

Implantation surgery Surgery will be performed by Jonathan Cheng, MD, at Clements University Hospital at UT Southwestern Medical Center in Dallas. Another staff hand surgeon or a hand surgery fellow or plastic surgery resident trainee may accompany him as an assistant during the procedure. General anesthesia will be provided by the Department of Anesthesiology at UT Southwestern. Procedures are estimated to last 4-6 hours, and will require placement of a standard catheter for intravenous (IV) access and a urethral (Foley) catheter for urine output monitoring. Long-lasting neuromuscular blockade will be avoided in the anesthetic regimen, in order to permit neuromuscular microstimulation / nerve conduction to help confirm neural anatomy during the surgical procedure. Preoperative IV antibiotic will be administered for infection prophylaxis. One 4-6 inch-long incision will be needed for implantation of nerve electrodes. The implant lead wires will be tunneled under the skin for a distance, and then placed through the skin. In the forearm-level amputees the wire exit sites may be below or above the elbow depending on the subject's prosthesis configuration. In the arm-level amputees the wire exit sites may be below or above the shoulder depending on the subject's prosthesis configuration. Small counter incisions may be needed along the paths of the lead wires to facilitate placement. The point where the lead wires exit the skin will be dressed with a sterile/antimicrobial dressing used commonly for indwelling vascular access devices (VAD). Following implantation, incisions will be infiltrated with bupivacaine for postoperative analgesia and closed with sutures and skin glue. The limb will be placed in a protective splint / immobilizer for the first 3 weeks after surgery.

Motor and somatosensory evoked potentials Nerve dissection will be performed under the operating microscope or surgical loupes. The motor and sensory fascicular groups of the ulnar and median nerves will be identified microsurgically as needed for the planned electrode implantations (ulnar only, or ulnar+median) based on their predictable intraneural topography.

Nerve electrode implantation The ulnar and median nerves will be accessed through a skin incision (4-6 inches long). The nerves will be microdissected with 2 electrode arrays targeted to the component fascicles of the ulnar nerve and 2-5 electrode arrays to the component fascicles of the median nerve.

Post-operative care in the hospital Immediately following surgery, subjects will receive routine postoperative care. Overnight hospital stay for up to 2 nights will be optional depending on the level of pain control in the PACU following surgery. Analgesia will consist of acetaminophen and parenteral and oral narcotics, and pregabalin or gabapentin and/or nortriptyline as needed for neuropathic pain. The Foley catheter will be removed as soon as possible following surgery. The IV fluids will be capped as soon as the patient demonstrates adequate oral intake and normal fluid balance. The patient will wear sequential devices on the legs and will walk on a scheduled basis for venous thromboembolism prophylaxis. Prophylactic antibiotics will be administered during the hospital stay up to 24 hours after surgery. Discharge criteria will be met when the patient demonstrates pain controlled adequately by oral analgesics, independent ambulation, and tolerance of oral intake.

X-rays After implantation surgery, plain film x-rays will be obtained of the subject's limb in order to establish a baseline for the position of implanted electrodes and leads.

Outpatient care The subject will be seen in clinic on a weekly basis following implantation surgery for 3 weeks and then as needed until explantation if there is evidence of local redness, inflammation, serous drainage or skin irritation near the incisions.

Percutaneous leads The electrode leads will be inspected at each weekly visit, and the dressings will be changed using sterile technique based on VAD protocols. If any dressing ever becomes wet, soiled, or leaking, the subject will be instructed to change it. After the first 3 clinic visits wire site dressing changes will be performed by research personnel who have been trained by the principal investigator.

Experimental data collection in implanted subjects (2 - 540 +/- 30 days)

Timing: Human physiology experiments will begin after 2 days following implantation, to allow tissue-electrode interactions to stabilize. Subjects will have human physiology lab sessions up to 6 times per month.

Location: Most of the human physiology experiments will take place at UT Southwestern. Some participants may be asked to travel to the University of Minnesota Bioengineering Lab up to 10 times during the study participation period for the human physiology experiments. Subjects also may be asked to participate in experimental sessions outside of the laboratory, in order to measure the impact of non-laboratory environmental settings on nerve recordings and subject perception of sensory nerve stimulation. These will take place in a controlled environment, supervised by member(s) of the research team during experimental trials, which may include a clinical exam room or therapy space, conference or meeting room, hotel room or private residence. These sessions may take place one time a month, for up to 7 days at a time.

Motor assessment: We will ask subjects to attempt to perform hand movements and positions. The movement trials will consist of simultaneous volitional movements and positioning of both the uninjured/sound limb and the injured/amputated "phantom" limb. We will record nerve electrode activity during all of the movement trials.

Sensory assessment: We will also perform sensory detection and discrimination trials. Here, the subject will be asked to report if he/she detects any sensation during microstimulation via implanted electrodes. If they do have a sensory perception, they will be asked to describe the quality and strength of the perception, e.g. location, touch, vibration, temperature. Subjects may also be asked to fill out standardized sensory/pain assessments during microstimulation and after microstimulation is turned off. Other stimulation trials that may be done will include single or multiple electrode stimulation to see if subjects can perceive multiple sensory percepts simultaneously.

Sensory-motor integration: After determining the subject's sensory detection and discrimination parameters, we will ask them to perform activities using the prosthetic hand. Microstimulation via implanted electrodes will be paired with motion or contact during task performance in order to determine whether providing evoked sensation during prosthesis use improves task-based performance.

Autonomic assessment: Noninvasive studies maybe performed up to 6 times to assess normal body functions reflecting the activity of the autonomic nervous system, such as EKG (electrocardiogram), temperature, heart rate, pulse oximetry, blood pressure, cutaneous sweat production, and cutaneous blood flow using laser Doppler.

Explantation surgery - Will be planned for 540 +/- 30 days after implantation. If explantation surgery is scheduled for less than 90 days from the implantation pre-operative testing then the pre-operative testing requirement will be waived. Surgery will be performed by the PI. General anesthesia will be provided by the Department of Anesthesiology at UT Southwestern. Procedures are estimated to last 2-3 hours, and will require placement of a standard catheter for IV access. Preoperative IV antibiotic will be administered for infection prophylaxis. The previous incisions used to place nerve electrodes will be redeveloped for access to the implanted systems. Following explantation, incisions will be infiltrated with bupivacaine for postoperative analgesia and closed with sutures and skin glue. Postoperative analgesia will be performed as listed above. Jonathan Cheng, MD, will see the subject in clinic once the week following surgery and then as needed. The dressing will be removed and replaced at the first postoperative visit. The incisions will be visually inspected at each visit. The subject will be instructed to contact the research team by phone on week 2 and week 3 to determine if they need to come to the clinic.

Post-participation interview - Subjects may be asked to participate in a recorded video interview conducted by the research team to record their subjective experiences with the study.

ELIGIBILITY:
Criteria for Inclusion of Subjects:

Hand, forearm and arm amputees:

1. Male or female, age 18 and older, of any race or ethnicity
2. Able and willing to sign Consent
3. Able and willing to participate in all study activities including implantation, testing and explantation of the study device.
4. Able to communicate effectively in English without an interpreter

After preliminary screening subjects will be assessed for the following inclusion criteria:

Overall and phantom pain are well-controlled and not incapacitating

Criteria for Exclusion of Subjects:

1. If MR neurogram and EMG/NCS study show nerve or muscle dysfunction/injury at a higher level than anticipated based on the appearance of the physical amputation stump, the subject may be excluded from the study due to adverse neuromuscular anatomy which would preclude use of the proposed experimental electrode implants. The radiographs will be used to confirm suitability of the amputation stump configuration. If the bony anatomy of the amputation stump is found to be unsuitable, the patient may be excluded from the study.
2. Subjects who have a history of cardiac arrhythmia will be excluded from the study.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-06; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Motor Assessment | up to 6 times per month beginning 2 days after implantation up to day 540 +/- 30 days
  We will ask you to attempt to perform hand movements and positions. The movement trials will consist of simultaneous volitional movements and positioning of both the uninjured/sound limb and the injured/amputated "phantom" limb done. This allows us to have a physical record of exactly what movement is being attempted by the amputated limb. We will record nerve and muscle electrode activity during all of the movement trials. During some movement trials, we will stimulate the LIFE neural electrodes while recording from implanted vs. surface adhesive vs. percutaneous needle muscle electrodes
Sensory Assessment | up to 6 times per month beginning 2 days after implantation up to day 540 +/- 30 days
  We will also perform sensory detection and discrimination trials. Here, you will be asked to report if you detect any sensation during microstimulation (delivering very small electrical signals) via LIFE electrodes. If you do have a sensory perception, you will be asked to describe the quality and strength of the perception, e.g. location, touch, vibration, temperature. You may also be asked to fill out standardized sensory/pain assessments during microstimulation and after microstimulation is turned off. Other stimulation trials that may be done will include single or multiple electrode stimulation to see if subjects can perceive multiple sensory percepts simultaneously. Blinded trials may be done to determine if the subjects are actually perceiving the same percept for a given stimulation paradigm. Other trials may include modulating the stimulation parameters to determine if the sensory percept changes characteristics with varying stimulation paradigms.
Sensory-Motor Integration | up to 6 times per month beginning 2 days after implantation up to day 540 +/- 30 days
  After determining your sensory detection and discrimination parameters, we will ask you to repeat standardized assessments using the existing myoelectric partial hand prosthesis. Microstimulation via LIFE electrodes will be paired with motion or contact during task performance in order to determine whether providing evokes sensation during prosthesis use improves task-based performance.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Cheng, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen AT, Drealan MW, Khue Luu D, Jiang M, Xu J, Cheng J, Zhao Q, Keefer EW, Yang Z. A portable, self-contained neuroprosthetic hand with deep learning-based finger control. J Neural Eng. 2021 Oct 11;18(5). doi: 10.1088/1741-2552/ac2a8d. PMID 34571503
- [Derived] Nguyen AT, Xu J, Jiang M, Luu DK, Wu T, Tam WK, Zhao W, Drealan MW, Overstreet CK, Zhao Q, Cheng J, Keefer EW, Yang Z. A bioelectric neural interface towards intuitive prosthetic control for amputees. J Neural Eng. 2020 Nov 11;17(6). doi: 10.1088/1741-2552/abc3d3. PMID 33091891
- [Derived] Overstreet CK, Cheng J, Keefer EW. Fascicle specific targeting for selective peripheral nerve stimulation. J Neural Eng. 2019 Nov 11;16(6):066040. doi: 10.1088/1741-2552/ab4370. PMID 31509815